CLINICAL TRIAL: NCT05519254
Title: Lactoferrin and Lysozyme Supplementation for Long-term Diarrhea Sequelae
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Patricia B Pavlinac, Associate Professor, SPH: Global Health, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00011759; 1R01HD103642-01 (NIH)
Record Dates: First submitted 2022-08-03; First posted 2022-08-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Diarrhea; Wasting; Malnutrition, Child
MeSH Terms: conditions — Diarrhea; Cachexia; Child Nutrition Disorders | interventions — Lactoferrin; Muramidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lactoferrin Arm (Experimental): 16-week course of lactoferrin
  Interventions: Dietary Supplement: Lactoferrin
- Lysozyme Arm (Experimental): 16-week course of lysozyme
  Interventions: Dietary Supplement: Lysozyme
- Combination Arm (Lactoferrin + Lysozyme) (Experimental): 16-week course of lactoferrin and lysozyme
  Interventions: Combination Product: Lactoferrin + Lysozyme
- Placebo Arm (Placebo Comparator): 16-week course of taste/appearance-matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactoferrin — Caregivers of children will be instructed to provide 1.5g of lactoferrin with 40g of unmodified rice powder daily mixed with 125 mL of porridge or other complimentary food.
  Arms: Lactoferrin Arm
Dietary Supplement: Lysozyme — Caregivers of children will be instructed to provide 41.5g of Lysosure daily mixed with 125 mL of porridge or other complimentary food.
  Arms: Lysozyme Arm
Combination Product: Lactoferrin + Lysozyme — Caregivers of children will be instructed to provide 40g of Lysosure with 1.5 grams of lactoferrin daily mixed with 125 mL of porridge or other complimentary food.
  Arms: Combination Arm (Lactoferrin + Lysozyme)
Other: Placebo — Caregivers of children will be instructed to provide 41.5 grams of unmodified rice powder daily mixed with 125 mL of porridge or other complimentary food.
  Arms: Placebo Arm

SUMMARY:
Children in low- and middle-income countries who are hospitalized for diarrhea and also have malnutrition are at high risk for illness and death in the 6 months period following treatment for diarrhoea despite receiving current guideline recommended diarrhea management (such as oral rehydration solution, or "ORS"). This study will test whether nutritional supplements made from milk (lactoferrin or lysozyme) or a combination of the two (lactoferrin and lysozyme) will prevent children from having repeated diarrhea episodes and help improve their nutrition by improving their stomach health or preventing new disease during this 6-month period. The study is taking place at 7 hospitals in Western Kenya. Six hundred participants will be enrolled if they provide informed consent to participate, are aged 6-24 months, were hospitalized with diarrhea and malnutrition and have been managed by the facility nutritionists and ready to return home. Participation in the study will entail providing information on the child's health history, collection of stool samples, blood, and potentially urine. The caregiver will be provided sachets of the investigational product to take home and mix daily with their child's porridge or other complimentary food, and asked to return to the clinic 4 times in the subsequent 6 months, and also consent to having a community health worker visit their home every two weeks for a follow up visit. The risks to the participant and their caregiver are minimal. The information gained in this study will help us create new treatments and develop new strategies to treat sick children to prevent death and illness.

DETAILED DESCRIPTION:
Current diarrhea management strategies in low- and middle-income countries (oral rehydration solution, ReSoMal and zinc) focus primarily on the management of dehydration and micronutrient replacement and appear to have negligible impact in preventing future diarrheal episodes or improving nutritional outcomes. Lactoferrin and lysozyme are milk-derived nutritional supplements that may reduce the risk of diarrheal episodes and accelerate nutritional recovery by treating or preventing underlying enteric infections and/or improving enteric function. Children with moderate or severe wasting are at particularly high-risk of death, diarrhea recurrence, and nutritional deterioration following a diarrheal episode. This factorial, double-blind, placebo-controlled, randomized trial aims to determine the efficacy of lactoferrin and lysozyme supplementation in decreasing diarrhea incidence and improving nutritional recovery in children convalescing from diarrhea and wasting. We will explore whether these interventions improve outcomes by reducing enteric pathogens, improving enteric function and/or increasing hemoglobin concentrations in these children. This study aims to enroll 600 Kenyan children aged 6-24 months from facilities in Western Kenya. Enrolled children will be randomized to 16-weeks of lactoferrin, lysozyme, a combination of the two, or placebo and be followed up for 24 weeks total, with bi-weekly home visits by community health workers and clinic visits at 4, 10, 16, and 24 weeks. Results of this study will inform management strategies for children with moderate/severe wasting at high risk for mortality, morbidity, and nutritional deterioration following diarrhea.

Aim 1: To determine whether a 16-week course of lactoferrin, lysozyme or a combination of both shortens time to WHO-defined recovery from wasting (MUAC ≥12.5cm) and reduces the incidence of moderate-to-severe diarrhea during the subsequent 6-months following presentation to a health facility with diarrhea among children with moderate/severe childhood wasting (MUAC <12.5 cm at the time of screening).

Hypothesis: Children randomized to lactoferrin, lysozyme, or the combination of both will experience a lower incidence of moderate-to-severe diarrhea and an earlier recovery from wasting (increased MUAC) over the subsequent 6-months than placebo-treated children. Combination therapy will provide synergistic benefit in reducing diarrhea and improving nutritional recovery.

Aim 2: To explore whether a 16-week course of lactoferrin, lysozyme or combination therapy improves secondary clinical, nutritional, enteric pathogen, and enteric function outcomes.

Hypothesis: Children randomized to lactoferrin, lysozyme, or the combination will experience fewer hospitalizations and deaths, improved linear growth, a reduced prevalence of specific enteric bacteria associated with linear growth failure (Campylobacter, LT-ETEC, EAEC, typical EPEC and/or Shigella), improved markers of enteric dysfunction (myeloperoxidase, alpha antitrypsin, neopterin, and the lactulose:rhamnose ratio) and improved hemoglobin, as compared to placebo-treated children.

Aim 3: To evaluate acceptability, adherence and cost-effectiveness of lactoferrin and/or lysozyme in Kenya.

Hypothesis: Both therapies will be highly acceptable to caregivers and health workers. Adherence to the therapies will be high among participants (≥ 95%). Lactoferrin and lysozyme, alone and in combination, will be more cost-effective interventions for reducing moderate-to-severe diarrhea in the short-term as compared to the standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-24 months
* Managed as an outpatient or inpatient for diarrhea at one of the recruiting sites
* MUAC <12.5 cm at the time of screening
* Plan to stay within the study area for the next 6 months or greater

Exclusion Criteria:

* Age younger than 6 months or older than 24 months
* Caregiver does not provide consent to study participation
* History of 2 or more blood transfusions in the past 12 months
* Exclusively breastfeeding at the time of enrollment
* History of congenital defect or syndrome that prevents age-appropriate feeding (e.g. cleft palate)
* History of allergy to dairy products
* Child is not ready to return home (is not yet discharged), or discharged against medical advice
* Unwilling to participate in the dual sugar permeability sub-study if selected
* Enrollment in another study

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate-to-severe diarrhea | 6 months
  Defined as total number of new diarrhea episodes (> 48 hours after a diarrhea-free period) deemed moderate-to-severe, divided by the child-time at risk during the 6-month follow-up period. Moderate-to-severe diarrhea will be defined as ≥ 3 using the CODA (Community DiarrhoeA) diarrhea severity score or dysentery (evidence or reported visible blood in stool).
Time to nutritional recovery | 6 months
  Defined as the number of days since enrollment to the date of the second of two consecutive MUAC measurements ≥ 12.5 cm.

SECONDARY OUTCOMES:
Incidence of diarrhea (any severity) | 6 months
  Diarrhea (any severity) will be defined as diarrhea (3 or more abnormally loose or watery stool) during follow-up, irrespective of severity, ascertained through follow-up visit questionnaires and a diarrhea diary. Episodes will be defined as per the primary outcome.
Incidence of severe diarrhea | 6 months
  Severe diarrhea defined by the CODA diarrhea severity score of 7 or more or dysentery. Episodes will be defined as per the primary outcome.
Incidence of dysentery | 6 months
  Dysentery will be defined as evidence or reported visible blood in stool. Episodes will be defined as per the primary outcome.
Incidence of medically-attended diarrhea | 6 months
  Medically-attended diarrhea will be defined as diarrhea that led to an outpatient or inpatient visit at a health facility or hospital that is typically attended by a nurse, clinical officer, and/or physician. Episodes will be defined as per the primary outcome.
Cumulative duration of diarrhea | 6 months
  Defined as cumulative days of diarrhea ascertained from follow-up visit questionnaires and a diarrhea diary, irrespective of episodes
Proportion of children who recovered from wasting based on two consecutive MUAC measurements ≥12.5 at any point during the follow-up period. | 6 months
Incidence of hospitalization | 6 months
  Defined as any inpatient admission that results in an overnight stay (irrespective of diagnosis) in a health-facility and time to hospitalization or death analyzed as a combined outcome
Composite outcome of time to hospitalization and death | 6 months
  Hospitalization will be defined as any inpatient admission that results in an overnight stay (irrespective of diagnosis) in a health-facility
Hemoglobin concentration | Measured at week 16
  Will be determined at week 16
Change in length for age z-score (linear growth) | 6 months
  Growth that includes length and weight measurements at each time point will be used to create age-standardized z-scores, calculated using WHO-established reference standards and the WHO ANTHRO software. Linear growth will be defined as change (Δ) in LAZ.
Change in weight for length z-score | 6 months
  Growth that includes length and weight measurements at each time point will be used to create age-standardized z-scores, calculated using WHO-established reference standards and the WHO ANTHRO software. Ponderal growth will be defined as change (Δ) in weight for length z-score (WLZ) and Δ MUAC.
Change in mid-upper arm circumference (cm) | 6 months
  Growth that includes length and weight measurements at each time point will be used to create age-standardized z-scores, calculated using WHO-established reference standards and the WHO ANTHRO software. Ponderal growth will be defined as change (Δ) in weight for length z-score (WLZ) and Δ MUAC.
Concentration of fecal alpha antitrypsin (mg/g) | Measured at baseline, week 4, 16, and 24
  Fecal biomarker of enteric function
Concentration of fecal myeloperoxidase (ng/mL) | Measured at baseline, week 4, 16, and 24
  Fecal biomarker of enteric function
Concentration of fecal calprotectin (mcg/g) | Measured at baseline, week 4, 16, and 24
  Fecal biomarker of enteric function
Lactulose:rhamnose ratio | Measured at week 4, 10, 16, and 24 for a subset of 200 participants (50 per arm)
  Lactulose:rhamnose ratio is a functional assessment of enteric integrity. Ratio will be measured in subset of 50 children per arm (200 children total).
Proportion of participants with enteric infections | Measured at week 4 for all participants and at week 16 and 24 for a subset of 200 participants (50 per arm)
  Determined by qPCR at or below the minimum limit of detection (cycle thresholds [CT] <35)
Proportion of caregivers reporting that administration of lactoferrin and/or lysozyme was desirable or satisfactory via 5-point Likert scale responses in surveys and focus group discussions (FGDs) | Week 4, 10, 16 (surveys) and 6 months (FGDs)
  Acceptability measure
Proportion of caregivers reporting perceived trust, safety, and comfort in administering lactoferrin and/or lysozyme via 5-point Likert scale responses in surveys and focus group discussions (FGDs) | Week 16 (surveys) and 6 months (FGDs)
  Acceptability measure
Proportion of caregivers self-reporting their child consumed some or all of the investigational product ≥95% of the time using daily pictorial logs | 16 weeks
  Adherence measure
Proportion of children adherent to the recommended dosing based on objectively measured container consumption (± 10% consumption of prescribed IP in all weeks) | 16 weeks
  Adherence measure
Incremental costs of diarrhea | 6 months
  Incremental costs of diarrhea will be measured in each arm and compared to the placebo arm
Cost-per-episode of diarrhea averted | 6 months
  Cost-per-episode of diarrhea averted will be measured in each arm and compared to the placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Patricia B Pavlinac, Principal Investigator — University of Washington
Locations (4):
- Kenya (4):
  - Homa Bay County Referral Hospital, Homa Bay
  - Isebania Sub-County Hospital, Isibania
  - Kisii Teaching and Referral Hospital, Kisii
  - Rongo Sub-County Hospital, Rongo

IPD SHARING:
Plan to Share IPD: Yes
The de-identified analytic dataset and analytic R code will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication.
Access Criteria: Publicly available

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Tickell KD, Pavlinac PB, John-Stewart GC, Denno DM, Richardson BA, Naulikha JM, Kirera RK, Swierczewski BE, Singa BO, Walson JL. Impact of Childhood Nutritional Status on Pathogen Prevalence and Severity of Acute Diarrhea. Am J Trop Med Hyg. 2017 Nov;97(5):1337-1344. doi: 10.4269/ajtmh.17-0139. PMID 29140236
- [Background] Talbert A, Ngari M, Bauni E, Mwangome M, Mturi N, Otiende M, Maitland K, Walson J, Berkley JA. Mortality after inpatient treatment for diarrhea in children: a cohort study. BMC Med. 2019 Jan 28;17(1):20. doi: 10.1186/s12916-019-1258-0. PMID 30686268
- [Background] Tickell KD, Sharmin R, Deichsel EL, Lamberti LM, Walson JL, Faruque ASG, Pavlinac PB, Kotloff KL, Chisti MJ. The effect of acute malnutrition on enteric pathogens, moderate-to-severe diarrhoea, and associated mortality in the Global Enteric Multicenter Study cohort: a post-hoc analysis. Lancet Glob Health. 2020 Feb;8(2):e215-e224. doi: 10.1016/S2214-109X(19)30498-X. PMID 31981554
- [Background] Brander RL, Pavlinac PB, Walson JL, John-Stewart GC, Weaver MR, Faruque ASG, Zaidi AKM, Sur D, Sow SO, Hossain MJ, Alonso PL, Breiman RF, Nasrin D, Nataro JP, Levine MM, Kotloff KL. Determinants of linear growth faltering among children with moderate-to-severe diarrhea in the Global Enteric Multicenter Study. BMC Med. 2019 Nov 25;17(1):214. doi: 10.1186/s12916-019-1441-3. PMID 31767012
- [Background] Cheng WD, Wold KJ, Bollinger LB, Ordiz MI, Shulman RJ, Maleta KM, Manary MJ, Trehan I. Supplementation With Lactoferrin and Lysozyme Ameliorates Environmental Enteric Dysfunction: A Double-Blind, Randomized, Placebo-Controlled Trial. Am J Gastroenterol. 2019 Apr;114(4):671-678. doi: 10.14309/ajg.0000000000000170. PMID 30829679
- [Background] Ochoa TJ, Chea-Woo E, Baiocchi N, Pecho I, Campos M, Prada A, Valdiviezo G, Lluque A, Lai D, Cleary TG. Randomized double-blind controlled trial of bovine lactoferrin for prevention of diarrhea in children. J Pediatr. 2013 Feb;162(2):349-56. doi: 10.1016/j.jpeds.2012.07.043. Epub 2012 Aug 30. PMID 22939927
- [Background] Zavaleta N, Figueroa D, Rivera J, Sanchez J, Alfaro S, Lonnerdal B. Efficacy of rice-based oral rehydration solution containing recombinant human lactoferrin and lysozyme in Peruvian children with acute diarrhea. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):258-64. doi: 10.1097/MPG.0b013e31802c41b7. PMID 17255841
- [Derived] Tiwari R, Tickell KD, Yoshioka E, Otieno J, Shah A, Richardson BA, Keter L, Okello M, Nyabinda C, Trehan I, McGrath CJ, Means AR, Houpt ER, Liu J, Platts-Mills JA, Njunge JM, Rwigi D, Diakhate MM, Nyaoke J, Ochola E, John-Stewart G, Walson JL, Pavlinac PB, Singa BO. Lactoferrin and lysozyme to promote nutritional, clinical and enteric recovery: a protocol for a factorial, blinded, placebo-controlled randomised trial among children with diarrhoea and malnutrition (the Boresha Afya trial). BMJ Open. 2024 Aug 9;14(8):e079448. doi: 10.1136/bmjopen-2023-079448. PMID 39122384

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT05519254/SAP_003.pdf
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05519254/ICF_001.pdf